CLINICAL TRIAL: NCT06064773
Title: Evaluation Of One Lung Ventilation With Ultrasound in Thorax Surgery Operations
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Hale Aksu, associate professor, Dokuz Eylul University
Other Study IDs: 2021/17-04
Record Dates: First submitted 2023-09-19; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: One Lung Ventilation
Keywords: One Lung Ventilation; Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: thoracic USG — the confirmation of double lumen tube placement with thoracic USG in thoracic surgery operations with one lung ventilation.

SUMMARY:
BACKGROUND: The aim of this study is to evaluate the confirmation of double lumen tube placement with thoracic Ultrasound (USG) in thorax surgery operations with one lung ventilation.

METHODS: In this prospective and observational study, 130 patients aged between 18-65 years in ASA (American Society of Anesthesiology) I-III risk class who will undergo thoracic surgery with the application of single-lung ventilation were included in the study. A double-lumen endobronchial tube was placed in the patients blindly. One-lung ventilation (OLV) was confirmed by thoracic USG by the anesthesiologist. The patient's demographic data, rapid clinical evaluation and USG data results, and intraoperative surgeon satisfaction were recorded.

DETAILED DESCRIPTION:
This prospective observational study was carried out in the Department of Anesthesiology and Reanimation, with the permission of the Ethics Committee of Dokuz Eylul University Medical Faculty Hospital (Ethics Committee Decision No:2021/17-04). Between 01.07.2021 and 01.12.2021, cases requiring single-lung ventilation by thoracic surgery in the operating room of Dokuz Eylul University Faculty of Medicine were included in the study.

Over 18 years old, patients who need OLV and undergoing elective surgery was determined as inclusion criteria. Furthermore patients did not want to participate in the study, with a narrowed trachea and/or a narrowed main bronchus that does not allow DLT placement, with endobronchial lesion in the main bronchus, with subcutaneous emphysema, having a chest tube due to pneumothorax, with pleural effusion, having a history of pleurodesis, bullous lung, patients with a history of tracheostomy and patients who will undergo emergency surgery determined as exclusion criteria for the study.

On the day of surgery, all patients were premedicated after a 20 G cannula was placed on the back of the hand before they were taken to the operating room. Routine anesthesia induction was performed after preoxygenation with 100% O2 for 5 minutes by monitoring 3-lead electrocardiography, peripheral oxygen saturation and noninvasive blood pressure in the patients who were taken to the operating room. After anesthesia induction, patients underwent double lumen tube intubation and after confirming single lung ventilation with thoracic USG (GE Healthcare LOGIQ e), tube location was confirmed by fiberoptic bronchoscopy (FOB) and clinical evaluation and recorded. Slip sign on USG was evaluated with M-mode imaging in the right and left lower quadrants of the thorax at the level of the costophrenic angles. When the bronchial lumen was clamped, the tube was considered to be positioned correctly if the left shift sign was selectively lost.

Age, gender, body mass index (BMI), AmericanSociety of Anesthesiologists score, co-morbidities (Hypertension, diabetes mellitus, malignancy, chronic obstructive pulmonary disease) duration of surgery, clinical and FOB evaluation results of the patients included in the study, in the supine position and in the lateral position during the intraoperative period. The determined DLT malpositions and the manipulations performed to correct them and the results of the evaluation with the thorax USG method, as well as the intraoperative surgeon satisfaction were recorded by the doctor who followed the case.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old, patients
* who need OLV and undergoing elective surgery

Exclusion Criteria:

* patients did not want to participate in the study,
* with a narrowed trachea and/or a narrowed main bronchus
* with endobronchial lesion in the main bronchus,
* with subcutaneous emphysema,
* having a chest tube due to pneumothorax,
* with pleural effusion,
* having a history of pleurodesis,
* bullous lung,
* patients with a history of tracheostomy
* patients who will undergo emergency surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Over 18 years old, patients who need OLV and undergoing elective surgery
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Thoracic USG sensitive and specificity values | immediatelay after the Replacement of double lumen ETT
  confirmation of DLT location with thorax USG in thoracic surgery operations in which Single Lung ventilation was applied, sensitive and specificity values

CONTACTS AND LOCATIONS:
Overall Officials: Hale Aksu, Principal Investigator — Associated prof
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
If researchers ask for share then will be decided

REFERENCES:
- [Result] Kanavitoon S, Raksamani K, Troy MP, Suphathamwit A, Thongcharoen P, Suksompong S, Oh SS. Lung ultrasound is non-inferior to bronchoscopy for confirmation of double-lumen endotracheal tube positioning: a randomized controlled noninferiority study. BMC Anesthesiol. 2022 May 30;22(1):168. doi: 10.1186/s12871-022-01707-4. PMID 35637457